## Creating a Sustainable Infrastructure for SARS-COV-2 Testing at Syringe Exchange Programs

Statistical Analysis Plan

Version date: 04/06/2023

NCT 04852848

## **Statistical Analysis Plan**

We examined intervention effects on COVID-19 testing rates immediately following the intervention, at 1-month follow-up, and at 2-month follow-up using contingency table analyses and reported Pearson  $\chi 2$  test statistics and odds ratios (ORs) as a measure of effect size.